CLINICAL TRIAL: NCT02401360
Title: A Controlled Study to Assess Clinical Gingivitis and Microbiome Following the Use of Multiple Oral Hygiene Products
Brief Title: A Study to Assess Clinical Gingivitis and Microbiome Following the Use of Multiple Oral Hygiene Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012135
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Dental Plaque; Dental Gingivitis
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Oral care regimen
  Interventions: Drug: China Crest® Pro-health 7 Complete Toothpaste
- Control Group (Placebo Comparator): Toothbrush and toothpaste
  Interventions: Drug: China Crest® Cavity Protection Toothpaste

INTERVENTIONS:
Drug: China Crest® Pro-health 7 Complete Toothpaste — Crest® pro-health manual toothbrush Crest® pro-health gum protection rinse
  Arms: Experimental Group
Drug: China Crest® Cavity Protection Toothpaste — Crest® meliliangje manual toothbrush
  Arms: Control Group

SUMMARY:
This study assessed the efficacy of an oral hygiene regimen relative to a standard marketed toothpaste and manual toothbrush.

ELIGIBILITY:
Inclusion Criteria:

* give written informed consent prior to their participation;
* be 18 to 65 years of age at the time of enrollment;
* agree not to participate in any other oral/dental product studies;
* agree to delay any elective dentistry (including a dental prophylaxis);
* agree to refrain from the use of any non-study oral care products (including floss and mouthrinse) during the course of the study;
* agree to return for the scheduled visits and follow study procedures;
* be in good general health as determined by the investigator/designee based on a review of the health history/update for participation in the study;
* have more than 10 bleeding sites at visits 1-3
* Consistency of bleeding site number at baseline may be considered;
* have a minimum of 18 natural teeth with facial and lingual scorable surfaces; and
* refrain from performing any oral hygiene or consuming anything by mouth (except a small amount of water) at least 4 hours prior to their appointment.

Exclusion Criteria:

* teeth that are grossly carious, fully crowned, extensively restored and have heavy dental calculus
* antibiotic, anti-inflammatory or anti-coagulant therapy within two weeks of to the baseline exam
* medical conditions that the investigator considers significant and that may compromise the evaluation of study results
* currently participating in any other clinical trial
* participated in a clinical trial for plaque/gingivitis within the previous 30 days
* pregnant or lactating
* orthodontic appliances or removable partial dentures
* soft or hard tissue tumor of the oral cavity
* advanced periodontal disease
* history of hepatitis, diabetes, or other communicable diseases
* history of rheumatic fever, heart murmur, mitral valve prolapse or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* history of significant adverse effects following the use of oral hygiene products such as toothpaste
* oral pathoses that could interfere with compliance and/or examinations or that need treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Gingivitis | Day 0
  Gingivitis was assessed according to the Gingival Bleeding Index
Gingivitis | Day 3
  Gingivitis was assessed according to the Gingival Bleeding Index
Gingivitis | Day 10
  Gingivitis was assessed according to the Gingival Bleeding Index
Gingivitis | Day 24
  Gingivitis was assessed according to the Gingival Bleeding Index

SECONDARY OUTCOMES:
Plaque Examination | Day 0
  The Modified Turesky Plaque Index was used to examine plaque.
Plaque Examination | Day 3
  The Modified Turesky Plaque Index was used to examine plaque.
Plaque Examination | Day 10
  The Modified Turesky Plaque Index was used to examine plaque.
Plaque Examination | Day 24
  The Modified Turesky Plaque Index was used to examine plaque.

CONTACTS AND LOCATIONS:
Overall Officials: Tao He, DDS, PhD, Principal Investigator — Procter and Gamble